CLINICAL TRIAL: NCT05656391
Title: Impact of Bread Diet on Intestinal Dysbiosis and Irritable Bowel Syndrome Symptoms in Quiescent Ulcerative Colitis: A Pilot Study
Brief Title: Impact of Bread Diet on Intestinal Dysbiosis and Irritable Bowel Syndrome Symptoms in Quiescent Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Principal Investigator, Xavier Aldeguer, Head of Gastroenterology Department, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RTC-2017-CU
Record Dates: First submitted 2022-12-01; First posted 2022-12-19 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Ulcerative Colitis in Remission

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment bread (Active Comparator): Dietary treatment consisted of daily consumption of 200 grams of bread produced following traditional breadmaking techniques
  Interventions: Dietary Supplement: Treatment vs control bread
- Control bread (Placebo Comparator): Dietary treatment consisted of daily consumption of 200 grams of bread produced following modern breadmaking techniques
  Interventions: Dietary Supplement: Treatment vs control bread

INTERVENTIONS:
Dietary Supplement: Treatment vs control bread — Consumption of 200 grams per day of either treatment or control bread for eight weeks

SUMMARY:
The present study aimed to compare the in vivo prebiotic properties of bread produced by traditional breadmaking techniques with that made using a modern breadmaking method on Irritable Bowel Syndrome-like symptoms in patients with quiescent Ulcerative Colitis. The expected outcome of the differential effects was a change in the faecal microbiome composition, which may indicate changes in the mucosa-associated microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ulcerative colitis according to established clinical and histological criteria as common clinical practice
* Remission of ulcerative colitis defined as a total Mayo score ≤2 and faecal calprotectin values under 250 ng/g
* Subjects aged over 18 years
* Moderate-to-severe IBS-like symptomatology defined by Rome IV criteria and IBS Symptom Severity Score (IBS-SSS) > 175.

Exclusion Criteria:

* Presence of flare-up of UC
* Coeliac disease, colectomy, or intestinal resection
* Antibiotic intake, prebiotic or probiotic treatment within 3 months before the study
* Any malignancy, pregnancy, or breastfeeding
* Intake of medication potentially influencing gastrointestinal function
* Disability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Changes in IBS-like symptomatology | Measurements were assessed at baseline (T0) and eight weeks (T1)
  Changes in IBS-like symptomatology were tested by IBS-Symptom Severity Score. The overall IBS-SSS score was calculated by totalling the punctuation of its five items. Each ranged from 0 to 100: (i) abdominal pain, (ii) number of days of abdominal pain during the last 10 days (number of days with abdominal pain x10), (ii) abdominal distension, (iv) satisfaction of defecatory behaviour, (v) interference of IBS symptoms in life. The possible range was then 0-500.

SECONDARY OUTCOMES:
Changes in the abundance of bacterial markers | Measurements were assessed at baseline (T0) and eight weeks (T1)
  Shifts of abundance of Eubacteria (EUB), A. municiphila (AKK), M. smithii (MSM), Bacteroidetes (BAC), Ruminococcus sp. (RUM), F. prausnitzii (FPRA) and E. coli (ECO) levels will be measured prior (T0) and after the intervention (T1). Results will be expressed as 16S gene copies of microbes per gram of faeces

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Aldeguer, Principal Investigator — Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (IdiBGi)
Locations (1):
- Hospital Doctor Josep Trueta, Girona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lluansi A, Lliros M, Carreras-Torres R, Bahi A, Capdevila M, Feliu A, Vila-Quintana L, Elias-Masiques N, Cueva E, Peries L, Torrealba L, Miquel-Cusachs JO, Sabat M, Busquets D, Lopez C, Delgado-Aros S, Garcia-Gil LJ, Elias I, Aldeguer X. Impact of bread diet on intestinal dysbiosis and irritable bowel syndrome symptoms in quiescent ulcerative colitis: A pilot study. PLoS One. 2024 Feb 16;19(2):e0297836. doi: 10.1371/journal.pone.0297836. eCollection 2024. PMID 38363772

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT05656391/Prot_SAP_000.pdf